CLINICAL TRIAL: NCT00467246
Title: The Use of a Long-Acting Sub-Cutaneous Insulin Analogue in the Management of Hyperglycaemic Emergencies
Brief Title: Sub-Cutaneous Insulin in Hyperglycaemic Emergencies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethics approval denied
Sponsor: The Royal Bournemouth Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIPI2
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2007-04-30 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes emergencies
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Levemir

SUMMARY:
Hyperglycaemic emergencies are associated with significant mortality (mortality in Diabetic Ketoacidosis 0.65 - 3.3% and in HyperOsmolar Non-Ketotic Coma 12 -17%). To reduce morbidity and mortality, prompt intervention and coma and close monitoring are essential. The study is designed to investigate whether a simple intervention with a long acting insulin can improve resolution of acidosis and hyperglycaemia, prevent recurrence of ketoacidosis and shorten hospital stay.

DETAILED DESCRIPTION:
This is a randomised trial concerning patients presenting in A & E with a diabetic emergency, either a Diabetic Ketoacidosis (DKA) or a Hyperosmolar Non-Ketotic Coma (HONC). Once informed consent has been given, each patient will receive standard intravenous treatment. They will also receive a daily sub-cutaneous bolus of either a long-acting insulin or a placebo.

Blood will be taken at regular intervals to analyse the rate of fall of glucose and normalisation of blood pH.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with a diabetic emergency aged 18 and above.

Exclusion Criteria:

* Patients who do not speak English and need a translator.
* Patients under the age of 18 years.
* Patients who are unable to give their consent and who do not have a relative present wiling to give assent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Time to normoglycaemia
Reduction of recurrence of ketoacidosis and hyperglycaemia.

SECONDARY OUTCOMES:
To investigate time to treatment in patients presenting with a hyperglycaemic emergency

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, MD, Principal Investigator — Royal Bournemouth Hospital; Martin Taylor, MD, Study Director — Royal Bournemouth Hospital